CLINICAL TRIAL: NCT00357578
Title: A Case Control Study of Age-Related Macular Degeneration (AMD) Examining Gene Expression Patterns in Circulating Monocytes From Peripheral Blood Samples
Brief Title: Genetic Study of Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000114; 00-EI-0114
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-19

CONDITIONS: Age-Related Macular Degeneration
Keywords: Macrophages; Biopsy; Genetic Analysis; Geographic Atrophy; Choroidal Neovascularization; Fibroblast; Disciform; Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy; Choroidal Neovascularization

SUMMARY:
This study will examine skin and blood cells for genetic changes related to the development of age-related macular degeneration, an eye disease that can significantly impair the ability to read, drive, and carry out daily activities. It is the most common cause of vision loss in people over the age of 50.

People with age-related macular degeneration and healthy normal volunteers age 50 years or older may be eligible for this study. Candidates will undergo a medical history, physical examination and eye examination with dilation of the pupils. Photographs of the eye will be taken with a special camera.

Study participants will have blood drawn three times (no more than 6 tablespoons each time) and will undergo three skin biopsies. For the skin biopsy, an anesthetic is injected under the skin and a small piece of skin-approximately 1/4-inch cube-is removed. The blood draws and biopsies will be done at 7- to 10-day intervals. In most cases, a single biopsy is done at each visit, but it may be necessary to take-at most-one additional biopsy from the other arm during the same visit. Patients will return for one follow-up visit 7 to 10 days after the last biopsy for examination of the biopsy site and removal of any stitches.

The results of this study may provide investigators information needed to develop new means of diagnosing and treating age-related macular degeneration.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) represents the most common cause of blindness in patients over the age of 50. While both hereditary and environmental factors appear to play a role in the pathogenesis of the disease, no common genetic mutations have been identified. This pilot study is intended to test the feasibility of evaluating the patterns of expression of genes that may be involved in the pathogenesis of AMD. The genes of interest are involved in the process of wound repair, cell injury and cell death. We hope to access the expression of these genes, but in tissues taken from non-ocular sites, in patients with AMD and in patients without AMD.

Biopsied skin fibroblasts and circulating monocytes from 62 patients will be obtained; 14 without AMD, 14 with at least one large (greater than 125 microns) druse, with geographic atrophy and/or choroidal neovascularization from AMD, 10 with geographic atrophy only, and 20 with choroidal neovascularization and/or disciform scar. The gene expression patterns from these tissues will be examined through various techniques including polymerase chain reaction, Northern blot analysis, differential display and microarray technology. The genetic expression patterns in patients with AMD will then be compared to age-matched control subjects. The primary outcome will be to determine the feasibility of obtaining skin and monocyte samples from patients with AMD, extracting RNA from these samples, and studying gene expression patterns. This study will provide investigators with information needed to develop subsequent studies of potential diagnostic tests.

ELIGIBILITY:
* INCLUSION CRITERIA:

INCLUSION CRITERIA 1 THROUGH 3 APPLY TO THE FIRST TWELVE PARTICIPANTS ENROLLED. INCLUSION CRITERIA 4 THROUGH 6 APPLY TO THE LAST 50 PARTICIPANTS ENROLLED.

1. AMD Patients: Diagnosis of AMD defined by the presence of at least one druse greater than 125 microns in diameter (4 patients) or geographic atrophy in at least one eye or choroidal neovascularization with drusen of any size in at least one eye (4 patients). (AMD cases only)
2. Age 60 years or older.
3. Age-matched control patients, absence of drusen or no more than 5 drusen less than 63 microns, absence of other diagnostic criteria for AMD, and age 60 years or older. The distribution of ages in the control group will be as similar as possible to the distribution of ages in the disease groups (4 patients).
4. AMD Patients: Diagnosis of AMD defined by the presence of at least one druse greater than 125 microns in diameter (10 patients), geographic atrophy (10 patients) and choroidal neovascularization with drusen of any size in at least one eye and/or disciform scar (20 patients). (AMD cases only) Presence of neovascularization and disciform scar formation will be verified by color photography.
5. Age 50 years or older.
6. Age-matched control patients: absence of drusen or no more than 5 drusen less than 63 microns, absence of other diagnostic criteria for AMD, and age 50 years or older. The distribution of ages in the control group.

EXCLUSION CRITERIA:

Patient age less than 50 years.

Presence of retinal disease involving the photoreceptors and/or outer retinal layers other than AMD loss such as high myopia, retinal dystrophies, central serous retinopathy, vein occlusion, diabetic retinopathy and uveitis or similar outer retinal diseases which have been present prior to the age of 50.

Opacities of the ocular media, limitations of pupillary dilation or other problems sufficient to preclude adequate stereo fundus photography.

Medical problems which make consistent follow-up over the treatment period unlikely (e.g., stroke, severe MI, terminal carcinoma).

Inability or inaccessibility to obtain dermal biopsy from the inner aspect of both arms due to previous trauma, underlying skin disorder which would preclude good wound healing, previous surgery of the arm or breast which could prevent good wound healing or induce other changes at the biopsy site.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-04-14; Study Completion 2007-09-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bird AC, Bressler NM, Bressler SB, Chisholm IH, Coscas G, Davis MD, de Jong PT, Klaver CC, Klein BE, Klein R, et al. An international classification and grading system for age-related maculopathy and age-related macular degeneration. The International ARM Epidemiological Study Group. Surv Ophthalmol. 1995 Mar-Apr;39(5):367-74. doi: 10.1016/s0039-6257(05)80092-x. PMID 7604360